CLINICAL TRIAL: NCT07363967
Title: A Phase I First-in-Human Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of SWA1211 Tablets in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing StoneWise Technology Co., Ltd (Industry)
Collaborators: Shanghai East Hospital (Other); Shanghai Cancer Centre (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWC0102
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation Study (Experimental): An accelerated titration design (ATD) combined with a traditional 3+3 dose escalation design of SWA1211 will be used. Six dose-escalation cohorts are planned.
  Interventions: Drug: SWA1211
- Phase 1b: Dose Expansion Study (Experimental): The trial will proceed to the dose expansion study after completion of dose escalation (Phase 1a) for SWA1211, with 1 to 2 cohorts, each with 20 ~ 30 subjects.
  Interventions: Drug: SWA1211

INTERVENTIONS:
Drug: SWA1211 — Planned doses administered orally as a tablet daily

SUMMARY:
The goal of this phase I, first-in-human, open-label study is to evaluate the safety, tolerability, PK, and preliminary anti-tumor activity of SWA1211 in subjects with advanced solid tumors. It includes a Phase Ia dose escalation study and a Phase Ib dose expansion study. The main questions it aims to answer are:

1. Assess the safety and tolerability of SWA1211 in subjects with advanced solid tumors.
2. Identify the dose-limiting toxicity (DLT) to establish the maximum tolerated dose (MTD) or maximum administered dose (MAD) and/or the recommended Phase II dose (RP2D) of SWA1211.
3. Assess the PK characteristics of SWA1211.
4. Evaluate the preliminary anti-tumor activity of SWA1211.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are fully informed of the purpose, nature, method, and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent document before any study procedure.
2. Subjects aged between 18 to 75 years old, male or female when signing the informed consent form (ICF).
3. Study population:

   Phase Ia (Dose Escalation Study): Subjects with histologically or cytologically confirmed advanced solid tumors, who have failed standard treatments, have no available standard treatment, or are not suitable for standard treatment at present.

   Phase Ib (Dose Expansion Study): Subjects with histologically or cytologically confirmed advanced solid tumors, who have failed standard treatments, have no available standard treatment, or are not suitable for standard treatment at present. The specific tumor types will be adjusted based on the results of Phase Ⅰa (dose escalation study).
4. Tumor tissue samples (preferable but not mandatory; fresh or archived) from patients will be collected during the screening period to assay the expression of HPK1. However, patient enrollment is not based on HPK1 expression levels.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of at least 3 months.
7. The function of bone marrow reserve and organs must meet the following requirements (without ongoing continuous supportive treatment):

   Bone marrow reserve: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 90 × 109/L, and hemoglobin (Hgb) ≥ 9.0 g/dL (no blood transfusion or hematopoietic stimulating factor therapy within 14 days).

   Coagulation function: Activated partial thromboplastin time (APTT) prolongation ≤ 1.5 × upper limit of normal (ULN), and international normalized ratio (INR) ≤ 1.5.

   Liver function: Total bilirubin (TBIL) ≤ 1.5 × ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (if there is liver metastasis, ALT or AST ≤ 5 × ULN).

   Kidney function: Creatinine clearance rate ≥ 60 mL/min (using the Cockcroft-Gault formula, see Appendix 1 for details); qualitative urine protein ≤ 1+, or qualitative urine protein ≥ 2+, but 24-hour urine protein < 1 g.

   Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; corrected QT interval (QTcF) ≤ 470 ms regardless of sex.
8. Subjects must have at least 1 evaluable lesion (only for Phase Ⅰa) or at least 1 measurable lesion (only for Phase Ⅰb) as defined by RECIST v1.1.
9. Eligible subjects with fertility (male and female) must agree to use reliable contraceptive methods (hormonal or barrier method or abstinence, etc., see Appendix 2 for details) with their partners during the study period and for at least 3 months after the last dose of the IP. For Female subjects of childbearing age, pregnancy test within 3 days before the first dose of IP must be negative.

Subjects who are able to communicate well with investigators, understand and adhere to the study requirements.

Exclusion Criteria:

1. Known to be allergic to SWA1211 tablets or any of their excipients (Polyvinyl caprolactam-polyvinyl acetate-polyethylene glycol graft copolymer; Vitamin E polyethylene glycol succinate, VE-TPGS 1000; Hypromellose; Propyl gallate; Methanol; Dichloromethane; Sodium lauryl sulfate; Microcrystalline cellulose; Manitol; Crospovidon; Silicon dioxide; Sodium stearyl fumarate; Film coating premix (Gastric dissolve type)).
2. Prior treatment with hematopoietic progenitor cell kinase 1 (HPK1) inhibitors.
3. Receipt of chemotherapy, radiotherapy, biological therapy, endocrine therapy, immune checkpoint inhibitor therapy, or other anti-tumor therapies within 4 weeks or 5 times the half-life of the drugs (whichever is longer) before the first dose of IP, except for the following items:

1)Have used nitrosourea or Mitomycin C within 6 weeks before the first dose of IP.

2)Have used oral fluorouracil and small molecule targeted drugs within 2 weeks or 5 times the half-life of the drugs before the first dose of IP (whichever is longer).

3)Have used herbal therapies with anti-tumor indications within 2 weeks before the first dose of IP.

4.Have received other clinical study drugs or treatments within 4 weeks before the first dose of IP, or still being within the safe follow-up period of other clinical study drugs or treatments.

5.Have received systemic glucocorticoids (> 10 mg/day of prednisone or equivalent), or other immunosuppressants within 14 days before the first dose of IP, with the following exceptions:

1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent).
2. Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption.
3. Short course (≤ 7 days) of corticosteroids prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by a contact allergen).

6.Use of CYP3A4 or CYP2C8 strong inducers or inhibitors within 14 days or 5 times the half-life of the drugs (whichever is longer) before the first dose of IP (see Appendix 3 for details).

7.Use of P-gp strong inhibitors, or P-gp substrates within 14 days or 5 times the half-life of the drugs (whichever is longer) before the first dose of IP (see Appendix 3 for details).

8.Use of acid-reducing agents (ARAs) (e.g., histamine H2-receptor antagonists (H2 blockers), and proton pump inhibitors (PPIs)) within 14 days or 5 times the half-life of the drugs (whichever is longer) before the first dose of IP.

9.Major organ surgery (excluding biopsy) or significant trauma or invasive dental procedures (such as tooth extraction, dental implants) within 4 weeks before the first dose of IP, or the requirement for elective surgery during the study period.

10.Have serious unhealable wounds, ulcers, or bone fractures within 4 weeks before the first dose of IP.

11.Bleeding events of grade 3 or above within 6 months before the first dose of IP, or currently ≥ grade 2 bleeding or factors judged by the investigator to have a high risk of bleeding (such as active peptic ulcer or esophageal varices) at present.

12.The adverse reactions of previous anti-tumor therapies have not yet recovered to ≤ grade 1 of CTCAE v5.0 (except for toxicities judged by the investigator to have no safety risk, such as hair loss, grade 2 peripheral neurotoxicity, etc.).

13.Have received immunotherapy and experienced ≥ grade 3 immune-related adverse events (irAEs), or ≥ grade 2 immune-related myocarditis.

14.Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence that such metastases have not been controlled, and the investigator judges it to be unsuitable for inclusion; 15.Gastrointestinal perforation, abdominal fistula, or intra-abdominal abscess occurred within 6 months before the first dose of IP, or the investigator has determined that there are high-risk factors for the formation of cavity organ perforation/fistula (such as tumor infiltration in the cavity Outer layer of the wall); inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis.

16.Unable to be dosed orally, or there are conditions judged by the investigator to seriously affect gastrointestinal absorption, such as dysphagia, uncontrolled nausea and vomiting, intestinal obstruction, chronic gastritis, gastroparesis syndrome, or gastric outlet obstruction.

17.Have active autoimmune conditions, or have a history of autoimmune diseases that may relapse (excluding well-controlled type 1 diabetes mellitus; manageable hypothyroidism with hormone replacement therapy only, or skin diseases that do not require systemic treatment, such as vitiligo or psoriasis).

18.Have active infection requiring systemic anti-infective treatment. 19.HIV infection, active HBV infection (with HBV DNA exceeding the ULN), or active HCV infection (with HCV RNA exceeding the ULN).

20.Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia that requires clinical intervention, or grade Ⅱ-Ⅲ atrioventricular block.
2. Thromboembolic events requiring therapeutic anticoagulation, or subjects with venous filters.
3. Subjects with grade III ~ IV cardiac insufficiency according to the New York Heart Association (NYHA) standards.
4. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other cardiovascular and cerebrovascular events of grade 3 or above occurring within 6 months before the first dose of the IP.
5. Clinically uncontrollable hypertension (where blood pressure cannot be controlled at systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg after standard antihypertensive treatment).
6. Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, or the use of any concomitant drugs known or suspected to prolong the QT interval.

21.Presence of clinically uncontrollable third-space effusion, as judged by the investigator.

22.History of interstitial lung disease (ILD) or evidence of history of pneumonitis on chest computed tomography scan within the 6 months before the first dose of the IP. Or interstitial lung disease that still requires glucocorticoid treatment at present (patients with radiation-induced pulmonary fibrosis not requiring hormone therapy are allowed to enroll).

23.Have a history of other malignant tumors within the 5 years before the first dose of the IP. However, patients with controlled basal cell carcinoma of the skin, cervical carcinoma in situ, breast carcinoma in situ, or squamous cell carcinoma of the skin may be enrolled.

24.Known history of drug abuse. 25.Presence of mental disorders or poor compliance. 26.Women who are pregnant or breastfeeding. 27.Inability to tolerate venous blood sampling. History of other serious systemic diseases, or other reasons judged by the investigator to make the subject unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose of study drug(s) to 90 days after the last dose or initiation of a new anticancer therapy, whichever occurs first; up to approximately 12 months
  1. Safety profile: adverse events (AEs, including irAEs), clinical laboratory tests (hematology, urinalysis, blood biochemistry, coagulation tests, cardiac enzymes, and cardiac troponin I (cTnI)), physical examination, vital signs, 12-lead electrocardiograms (12-lead ECG), ECOG, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided